CLINICAL TRIAL: NCT04814199
Title: Use of Standardized Algorithm for the Management of Epidural Analgesia for Labor and Delivery: An Observational Cohort Study
Brief Title: Use of Standardized Algorithm for the Management of Epidural Analgesia for Labor and Delivery
Status: Completed | Type: Observational
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 21-02
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2021-05

CONDITIONS: Labor Pain
Keywords: programmed intermittent epidural bolus; epidural analgesia; labor epidural
MeSH Terms: conditions — Labor Pain | interventions — Algorithms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients using epidural management algorithm: Patients will be educated and given an algorithm to follow while in labour and after having an epidural catheter placed.
  Interventions: Other: Algorithm

INTERVENTIONS:
Other: Algorithm — Patients will have a printed algorithm to follow while they are in labour with an epidural for pain management.
  Other Names: Epidural algorithm

SUMMARY:
Programmed Intermittent Epidural Bolus (PIEB) has become a standard technique for labour analgesia in many departments of anesthesia. Advantages to the former standard of care, continued epidural infusion (CEI), include reduced analgesic consumption , better maternal satisfaction and less occurrence of motor block . At Mount Sinai Hospital, the introduction of a bundle of changes in the management of labor analgesia including the use of PIEB, has resulted in an improvement of the quality of labor analgesia. This bundle of changes included labor catheter placement more often at L2/L3 interspace, more frequent use of fentanyl in the epidural loading dose, the implementation of a PIEB regimen and an increase in hourly baseline offer of local anesthetic.

A recent before-and-after study conducted by the investigators, comparing the current practice with the previous practice, which was based on CEI, identified that the incidence of women experiencing pain >3 (scale 0-10) (40% vs 30%) and the number of nurse-administered top-ups (24% vs 3%) were significantly reduced. However, despite that significant improvement, some 30% of women undergoing epidural analgesia still experience pain NRS >3 (NRS scale 0-10) during either first or second stage of labor.

Although the health care team attempts to manage epidurals as standardized as possible, there is some variation in practice resulting from the many stakeholders involved in the labor analgesia management, including anesthesiologists, obstetricians, nurses and patients. The investigators hypothesized that our most recent results may be explained by the lack of standardization of the management of epidural analgesia and that a standardized epidural catheter placement and a management algorithm may improve the efficacy of our epidural analgesia regimen.

The aim of this pilot study is to test the feasibility and efficacy of the use of a standardized algorithm for the management of labor epidural analgesia based on a PIEB regimen.

ELIGIBILITY:
Inclusion Criteria:

* request for epidural analgesia during labor
* ASA Physical Status II and III

Exclusion Criteria:

* patients requiring change in anesthetic management due to comorbidities or complications before initiation of epidural analgesia maintenance will be excluded.
* refusal to give written informed consent

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women admitted to the Labor and Delivery unit at Mount Sinai Hospital that request to receive epidural analgesia.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
Pain score, questionnaire | 24 hours
  Pain score using verbal numerical rating scale (VNRS) (0-10, where 0=no pain and 10=worst pain ever). This will be assessed hourly following epidural placement, as per institutional guidelines, until the patient delivers.
  The primary outcome of the study will be the presence of pain (NRS ≥ 3) at any time during the first and second stage of labor, after the establishment of an effective loading dose (pain NRS ≤ 1/10).

SECONDARY OUTCOMES:
Upper sensory block level | 24 hours
  The upper sensory block level to ice is defined as the dermatome at which there is an altered cold perception without complete sensitivity loss. This will be assessed hourly following epidural placement, as per institutional guidelines, until the patient delivers.
Motor block score using Bromage score | 24 hours
  Motor block will be assessed with the Bromage score: 0 = able to raise the extended leg; 1 = unable to raise the extended leg but able to flex knees; 2 = unable to flex knees, but able to flex ankle; 3 = unable to flex ankle. This will be assessed hourly following epidural placement, as per institutional guidelines, until the patient delivers.
Blood pressure | 24 hours
  Blood pressure measured hourly following epidural placement, as per institutional guidelines, until the patient delivers.
Heart rate | 24 hours
  Heart rate measured hourly following epidural placement, as per institutional guidelines, until the patient delivers.
Number of patient controlled epidural analgesia button presses | 24 hours
  Need for supplementary analgesia: the number of patient controlled epidural analgesia button presses will be recorded.
Number of top ups administered by nurses or physicians | 24 hours
  Need for supplementary analgesia: the number of top ups administered by nurses or physicians will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada